CLINICAL TRIAL: NCT06571201
Title: Patient-reported Outcomes and Esthetics With Single Dental Implants 10-15 Years After Placement, a Cross-sectional Study
Brief Title: Patient-reported Outcomes and Esthetics With Single Dental Implants
Status: Completed | Type: Observational
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Viveca Wallin Bengtsson, Prinicpal Investigator, phD, Kristianstad University
Other Study IDs: Single dental implants
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Patient Reported Outcome Measures; Patient Satisfaction; Implant Complication
Keywords: dental esthetics; patient reported outcome measurements; single dental implant
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate patient-reported long-term outcomes of single dental implants. Therefore, the aim of the study is to describe patient-reported functional and esthetic outcomes of single dental implants. A secondary aim is to evaluate the objective esthetics of single dental implants.

The primary outcomes are patient-reported experiences regarding the function, cleaning ability, and esthetics of the single dental implant. The esthetics of the single dental implant will also be assessed using the Pink Esthetic/White Esthetic Score Index and considered secondary outcome.

DETAILED DESCRIPTION:
Participants with one single-dental implant in the esthetic zone were selected. A clinical examination was performed and presence of bleeding (BOP), probing pocket depth (PPD) and presence of suppuration was registered. Two questionnaires with visual analogue scales (VAS) were filled in by the participants and intraoral photographs were taken. One of the questionnaires related to satisfaction with function and leaning and the other involved the esthetics of the single dental implant. One dentist reviewed the photographs using the pink esthetic score/white esthetic score (PES/WES) index.

Peri-implant mucositis was established if the presence of bleeding (BOP) and/or suppuration on gentle probing and the absence of bone loss beyond crestal bone level changes resulting from initial bone remodeling at the implant, according to the latest definition of Peri-Implant Diseases and Conditions. In this study, this was defined as ≤ 2.5 mm apical of the most coronal portion of the intra-osseous part of the implant.

A diagnosis of peri-implantitis was established if the presence of bleeding on gentle probing (BOP) and bone levels of ≥ 3 mm apical of the most coronal portion of the intra-osseous part of the implant, according to the latest classification of Peri-Implant Diseases and Conditions.

Parallel to medical records all data was saved in a safe together with a code list. The data was not opened until the study was completed and only by authorized persons with access to the data in the study such as, the principal investigator and the statisticians.

All participants was given oral and written information about the study and signed a written informed consent. The participants was informed that they could drop off whenever they wanted without any explanations. The ethical board approved the study and the investigation was performed according to the principles of the Declaration of Helsinki on experimentation involving human subjects.

The IBM SPSS version 28.0 statistical software package (SPSS Inc., Armonk, NY, USA) for personal computer was used in the statistical analyses. The data were analyzed using descriptive statistics with the mean and standard deviation (SD). Pearson's χ2 test and Mantel-Haenszel common odds ratios were used to analyze dichotomous data. For categorical data, percentages are given. Estimates (odds ratio, mean difference) are given with the corresponding 95% confidence interval. The significance level for the p value was set at 0.05. No data were missing. Cronbach's alpha was used to test the reproducibility of the PES/WES index used for the objective assessment of the esthetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* if only one single dental implant reconstruction in the esthetic zone, defined as teeth from the area of the upper right canine to the upper left canine
* if have filled in two questionnaires
* if answered an oral questionnaire
* if had intraoral photographs taken

Exclusion Criteria:

-if there was an edentulous area next to the implant to be studied

Ages: 23 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing prosthetic single dental implant treatment at an Oral Prosthodontic Specialist Clinic in Kristianstad (Folktandvården, Public Dental Service Kristianstad, Sweden) between 1991-1996
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-08-15 (Actual); Primary Completion 2007-06-07 (Actual); Study Completion 2007-06-07 (Actual)

PRIMARY OUTCOMES:
Patient- reported outcomes concerning function and cleaning of dental single implants | At the dental examination
  Visual Analogue Scale 0=yes absolutely 10= absolutely not. Maximum=100 scores Minimum=0 scores
Patient- reported outcomes concerning esthetics of dental single implants | At the dental examination
  Visual Analogue Scale 0=not satisfied at all. 10=completely satisfied Maximum=40 scores Minimum=0 scores

SECONDARY OUTCOMES:
Pink and white esthetic scores for single dental implants | 15 years later
  PES/WES index Belser et al. 2009 0=worst outcome and 2=best outcome reported by a dentist from intraoral photographs

CONTACTS AND LOCATIONS:
Overall Officials: Viveca Wallin Bengtsson, phD, Principal Investigator — University of Kristianstad
Locations (1):
- Kristianstad University, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gehrke P, Lobert M, Dhom G. Reproducibility of the pink esthetic score--rating soft tissue esthetics around single-implant restorations with regard to dental observer specialization. J Esthet Restor Dent. 2008;20(6):375-84; discussion 385. doi: 10.1111/j.1708-8240.2008.00212.x. PMID 19120783
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- [Background] Thoma DS, Cosyn J, Fickl S, Jensen SS, Jung RE, Raghoebar GM, Rocchietta I, Roccuzzo M, Sanz M, Sanz-Sanchez I, Scarlat P, Schou S, Stefanini M, Strasding M, Bertl K; working group 2 of the 6th EAO Consensus Conference 2021. Soft tissue management at implants: Summary and consensus statements of group 2. The 6th EAO Consensus Conference 2021. Clin Oral Implants Res. 2021 Oct;32 Suppl 21(Suppl 21):174-180. doi: 10.1111/clr.13798. PMID 34145925
- [Background] Altay MA, Sindel A, Tezerisener HA, Yildirimyan N, Ozarslan MM. Esthetic evaluation of implant-supported single crowns: a comparison of objective and patient-reported outcomes. Int J Implant Dent. 2019 Jan 7;5(1):2. doi: 10.1186/s40729-018-0153-3. PMID 30613918
- [Background] Pjetursson BE, Karoussis I, Burgin W, Bragger U, Lang NP. Patients' satisfaction following implant therapy. A 10-year prospective cohort study. Clin Oral Implants Res. 2005 Apr;16(2):185-93. doi: 10.1111/j.1600-0501.2004.01094.x. PMID 15777328
- [Background] Stefanini M, Felice P, Mazzotti C, Mounssif I, Marzadori M, Zucchelli G. Esthetic evaluation and patient-centered outcomes in single-tooth implant rehabilitation in the esthetic area. Periodontol 2000. 2018 Jun;77(1):150-164. doi: 10.1111/prd.12215. Epub 2018 Feb 28. PMID 29493024